CLINICAL TRIAL: NCT01894269
Title: Chemoembolization With or Without Antiviral Therapy for Unresectable HBV-related Hepatocellular Carcinoma With Low HBV DNA Replication: Effectiveness and Safety. A Prospective and Randomized Clinical Trial
Brief Title: Chemoembolization With or Without Antiviral Therapy for Unresectable HBV-related HCC With Low HBV DNA Replication
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiang-Ming Lao, MD, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sysucc-HCC010
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Lamivudine; entecavir; halofantrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anti-viral treatment (Experimental): Oral antiviral drugs will be commenced after TACE. That is: Lamivudine 100mg once daily; or Entecavir 0.5mg once daily.
  Interventions: Drug: Lamivudine 100mg once daily; or Entecavir 0.5mg once daily.
- Control (No Intervention): No anti-viral therapy after TACE.

INTERVENTIONS:
Drug: Lamivudine 100mg once daily; or Entecavir 0.5mg once daily. — In experimental group, Lamivudine 100mg once daily; or Entecavir 0.5mg once daily will be commenced after TACE.
  Other Names: lamivudine 100 mg tablets (GlaxoSmithKline);; Entecavir 0.5mg tablets (Bristol-Myers Squibb)
  Arms: Anti-viral treatment

SUMMARY:
Although it is commonly accepted that antiviral therapy should be commenced before or during hepatocellular carcinoma (HCC) treatment if the patients have high viral loads and elevated ALT or total bilirubin values with signs of cirrhosis, the dilemma exists when HBV DNA and liver function (such as ALT, AST, TBIL) remains low level. Whether antiviral therapy make sense or not in these patients with no signs of hepatitis or high viral replication remains unclear, especially for the relatively advanced stage HCC patients receiving TACE. Thus, the investigators carried out this prospective control study to compare the survivals for patients after TACE between with or without antiviral therapy.

DETAILED DESCRIPTION:
In highly endemic areas, hepatitis B virus (HBV) infection plays a primary role in the etiology of HCC and is frequently observed in HCC patients. Patients with HBV-related HCC usually have a history of chronic HBV infection. Chemotherapy for other malignancies has been associated with HBV reactivation. Furthermore, in end stage liver disease due to HBV, levels of HBV replication have been correlated with liver function. For TACE, reports on HBV reactivation have been inconsistent. Some studies have demonstrated HBV reactivation, some have not , and others have shown decreased HBV DNA levels . The exact mechanism by which this occurs is still unknown. Although anti-HBV therapy has been reported to suppress HBV reactivation in various clinical settings with immunosuppressive conditions, few reports were concerned with the TACE treatment of HBV-related HCC. Also, the long-term effects of antiviral therapy in relatively advanced HCC patients after HCC remains unclear.

Although it is commonly accepted that antiviral therapy should be commenced before or during HCC treatment if the patients have high viral loads and elevated ALT or total bilirubin values with signs of cirrhosis, the dilemma exists when HBV DNA and liver function (such as ALT, AST, TBIL) remains low level. Therefore, we would call for the establishment of clinical practice guidelines on the antiviral therapy in HBV-related HCC patients, especially a consensus on the indications to administer nucleosides analogs (NAs).

Thus , the purpose of the investigators' study is to prospectively study the efficacy of nucleosides analogs (NAs) in transcatheter arterial chemoembolization for nonresectable hepatocellular carcinoma with relatively low HBV DNA replication and Child-Pugh grade A based on multivariate analysis of prognostic factors. The HBV DNA and liver function parameters will be monitored closely. Once the reactivation occurs in the control group, antiviral therapy would be administered immediately. The study had a interim analysis to allow the trial to be stopped if significant differences were detected. The accumulated data were examined when half patient was enrolled in the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

Male or female patients from 18 to 75 years of age with a diagnosis of HCC. A diagnosis of HCC based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL).

The patient has not been previously treated with surgery, radiation therapy, radiofrequency ablation, percutaneous ethanol or acetic acid injection, or cryoablation, or any other treatment with chemotherapeutic agents or sorafenib.

The patient has not been previously treated with any anti-viral agents, including interferon or nucleosides analogs (NAs).

Adults patients with a diagnosis of HCC which is not amenable to surgical resection ,local ablative therapy or any other radically cured treatment.

The MDT group of HCC agree to administer TACE in this patient.

Patients must have at least one tumor lesion that can be accurately measured according to EASL criteria.

No serious concurrent medical illness.

Unresectable TNM stage Ⅲ or Ⅳ disease.

Zubrod-ECOG-WHO performance status: 0 or 1. and the estimated survival more than 4 months.

Not pregnant or breast-feeding patients

No significant renal impairment (creatinine clearance < 30 mL/minute) or patients on dialysis

No current infections requiring antibiotic therapy

Not on anticoagulation or suffering from a known bleeding disorder

No unstable coronary artery disease or recent MI

Ability to understand the protocol and to agree to and sign a written informed consent document

The following laboratory parameters at baseline:

Platelet count ≥ 70,000/µL

Hemoglobin ≥ 8.5 g/dL

Absolute neutrophil count (ANC) >1,500/mm3

Total bilirubin ≤ 1.5 mg/dL Serum albumin ≥ 35 g/L

Serum creatinine ≤ 1.5 x upper limit of normal

PT prolong time less than 3 seconds

Cirrhotic status of Child-Pugh class A only

ALT<2×upper limit of normal

Hepatitis B surface antigen positive

If hepatitis B e antigen positive, HBV DNA level <2000IU/mL; If hepatitis B e antigen negative, HBV-DNA<200IU/mL.

Exclusion Criteria:

- History of HIV or HCV infection.

History of organ allograft

Known or suspected allergy to the investigational agents or any agent given in association with this trial.

Evidence of bleeding diathesis.

Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.

Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of study entry.

Serious non-healing wound, ulcer, or bone fracture

Known central nervous system tumors including metastatic brain disease

Any event > grade 2 National Cancer Institute [NCI]-Common Terminology Criteria for Adverse Events [CTCAE] version 3.0

Severe complication after TACE.

History of hepatotoxic medication within 8 wk prior to the current treatment.

History of corticosteroid administration.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
overall survival | 1 year

SECONDARY OUTCOMES:
HBV reactivation | 1 year

OTHER OUTCOMES:
HBV resistance to lamivudine or entecavir | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jun Lin, MD, Principal Investigator — Sun Yat-sen University; Xiang-Ming Lao, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Yang HI, Lu SN, Liaw YF, You SL, Sun CA, Wang LY, Hsiao CK, Chen PJ, Chen DS, Chen CJ; Taiwan Community-Based Cancer Screening Project Group. Hepatitis B e antigen and the risk of hepatocellular carcinoma. N Engl J Med. 2002 Jul 18;347(3):168-74. doi: 10.1056/NEJMoa013215. PMID 12124405
- [Background] de Franchis R, Hadengue A, Lau G, Lavanchy D, Lok A, McIntyre N, Mele A, Paumgartner G, Pietrangelo A, Rodes J, Rosenberg W, Valla D; EASL Jury. EASL International Consensus Conference on Hepatitis B. 13-14 September, 2002 Geneva, Switzerland. Consensus statement (long version). J Hepatol. 2003;39 Suppl 1:S3-25. No abstract available. PMID 14708673
- [Background] Ho J, Wu PC, Kung TM. An autopsy study of hepatocellular carcinoma in Hong Kong. Pathology. 1981 Jul;13(3):409-16. doi: 10.3109/00313028109059059. PMID 6272177
- [Background] Lok AS, Lai CL, Wu PC, Wong VC, Yeoh EK, Lin HJ. Hepatitis B virus infection in Chinese families in Hong Kong. Am J Epidemiol. 1987 Sep;126(3):492-9. doi: 10.1093/oxfordjournals.aje.a114681. PMID 3618581
- [Background] Chen CJ, Yang HI, Su J, Jen CL, You SL, Lu SN, Huang GT, Iloeje UH; REVEAL-HBV Study Group. Risk of hepatocellular carcinoma across a biological gradient of serum hepatitis B virus DNA level. JAMA. 2006 Jan 4;295(1):65-73. doi: 10.1001/jama.295.1.65. PMID 16391218
- [Background] Liaw YF, Sung JJ, Chow WC, Farrell G, Lee CZ, Yuen H, Tanwandee T, Tao QM, Shue K, Keene ON, Dixon JS, Gray DF, Sabbat J; Cirrhosis Asian Lamivudine Multicentre Study Group. Lamivudine for patients with chronic hepatitis B and advanced liver disease. N Engl J Med. 2004 Oct 7;351(15):1521-31. doi: 10.1056/NEJMoa033364. PMID 15470215
- [Background] Shuqun C, Mengchao W, Han C, Feng S, Jiahe Y, Wenming C, Zhengfeng Y, Yuxiang Z, Peijun W. Antiviral therapy using lamivudine and thymosin alpha1 for hepatocellular carcinoma coexisting with chronic hepatitis B infection. Hepatogastroenterology. 2006 Mar-Apr;53(68):249-52. PMID 16608033
- [Background] Jang JW, Choi JY, Bae SH, Yoon SK, Chang UI, Kim CW, Cho SH, Han JY, Lee YS. A randomized controlled study of preemptive lamivudine in patients receiving transarterial chemo-lipiodolization. Hepatology. 2006 Feb;43(2):233-40. doi: 10.1002/hep.21024. PMID 16440357
- [Background] Piao CY, Fujioka S, Iwasaki Y, Fujio K, Kaneyoshi T, Araki Y, Hashimoto K, Senoh T, Terada R, Nishida T, Kobashi H, Sakaguchi K, Shiratori Y. Lamivudine treatment in patients with HBV-related hepatocellular carcinoma--using an untreated, matched control cohort. Acta Med Okayama. 2005 Oct;59(5):217-24. doi: 10.18926/AMO/31969. PMID 16286955
- [Background] Lao XM, Wang D, Shi M, Liu G, Li S, Guo R, Yuan Y, Chen M, Li J, Zhang Y, Lin X. Changes in hepatitis B virus DNA levels and liver function after transcatheter arterial chemoembolization of hepatocellular carcinoma. Hepatol Res. 2011 Jun;41(6):553-63. doi: 10.1111/j.1872-034X.2011.00796.x. Epub 2011 Mar 29. PMID 21615643
- [Background] Lao XM, Luo G, Ye LT, Luo C, Shi M, Wang D, Guo R, Chen M, Li S, Lin X, Yuan Y. Effects of antiviral therapy on hepatitis B virus reactivation and liver function after resection or chemoembolization for hepatocellular carcinoma. Liver Int. 2013 Apr;33(4):595-604. doi: 10.1111/liv.12112. Epub 2013 Feb 13. PMID 23402625
- [Background] Lao XM, Xia HH, Lin XJ, Li SP. Antiviral therapy in patients with hepatitis B virus-related hepatocellular carcinoma: is it ready for universal application? J Viral Hepat. 2013 Dec;20(12):e148-9. doi: 10.1111/jvh.12147. Epub 2013 Jul 17. No abstract available. PMID 24304460